CLINICAL TRIAL: NCT06852599
Title: Long-term Outcomes of Implants in Patients with Periodontitis
Acronym: Impl_longterm
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Dr. Antonio Ciardo, Principal Investigator, Heidelberg University
Other Study IDs: S-476/2023
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Peri-Implant Health; Periodontitis; Peri-implant Mucositis; Peri-implantitis
MeSH Terms: conditions — Periodontitis; Peri-Implantitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of the study is to examine potential influencing factors on the changes in the periodontal parameters probing pocket depth (PPD), bleeding on probing (BOP), and alveolar bone loss (ABL) on implants and control teeth (using a split-mouth design) over five (T-5), 7.5 (T-7), and ten years (T-10) of supportive periodontal care (SPC). For this purpose, 150 patients with periodontitis and implants are re-examined cross-sectionally (T0), and the changes in the main peri-implant and periodontal target parameters are compared retrospectively at the specified observation time points (T-5, T-7, T-10).

Potential influencing factors to peri-implant conditions include patient-related factors, therapy-related factors and implant-related factors. In addition, patients will be surveyed using validated questionnaires on oral health-related quality of life (OHIP-G14), and a number of common risk factors for periodontits and peri-implant conditions.

ELIGIBILITY:
Inclusion Criteria:

Patient-related:

* At least one dental implant present
* Age ≥ 18 years at the beginning of the observation period
* Verbal and written consent
* Complete periodontal and dental status at one of the defined observation time points with 6 probing sites per tooth/implant and bleeding on probing (BOP) recorded during the periodontal maintenance phase

Locally:

* a contralateral control tooth to the implant is present at the first defined observation time point
* BOP recorded on the implant

Exclusion Criteria:

* No written and verbal consent
* Younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study cohort is recruited from patients of the Department of Conservative Dentistry at Heidelberg University Hospital who have undergone systematic periodontal therapy, have a dental implant, and meet the other inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
changes in periodontal pocket depths | over five, 7.5, and ten years of supportive periodontal care

CONTACTS AND LOCATIONS:
Locations (1):
- Heidelberg University, Heidelberg, Baden-Wurttemberg, Germany